CLINICAL TRIAL: NCT00556517
Title: Acute Hamstring Strains in Danish Elite Soccer - Diagnosis and Biomechanical Tests
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Amager Hospital (Other)
Other Study IDs: H-A-2007-0063
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-09

CONDITIONS: Strains
Keywords: Hamstring; Strain; Rehabilitation; muscles
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A common soft tissue injury in sports involving sprinting and jumping is the hamstring strain. In addition to the frequency of injury, hamstring injuries are also the most recurrent soft tissue injury occurring in sport. There is a need for further research concerning diagnosis and different prognostic parameters for the rehabilitating process.

The aims for this study are:

A longitudinal comparison of sonographic and MRI assessments of acute and healing hamstring injuries.

A study investigating different biomechanical parameters in the process of determining whether a former hamstring injured soccer player is fully rehabilitated. We hypothesize that it is possible to use electromyography, muscle strength measurements and different tests on a force platform to help determine this issue.

ELIGIBILITY:
Inclusion Criteria:

* Acute hamstring strain caused during soccer activities (match or training)

Exclusion Criteria:

* A hamstring strain at the time for inclusion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male soccer players playing in one of the top 4 divisions in Denmark in the 2007/08 season.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-01; Study Completion 2009-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Petersen, MD, Principal Investigator — Department of Orthopaedic Surgery, Amager University Hospital, Denmark

REFERENCES:
- [Background] Petersen J, Holmich P. Evidence based prevention of hamstring injuries in sport. Br J Sports Med. 2005 Jun;39(6):319-23. doi: 10.1136/bjsm.2005.018549. PMID 15911599